CLINICAL TRIAL: NCT02262234
Title: Education Interventions for Self-Management of Pain Post-SCI: A Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: The Craig H. Neilsen Foundation (Other); Kessler Institute for Rehabilitation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-815-14
Record Dates: First submitted 2014-10-07; First posted 2014-10-13 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injury; Chronic Pain
Keywords: Spinal cord injury; Chronic pain; Education
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education Program Type 1 (Experimental)
  Interventions: Other: Education Program Type 1
- Education Program Type 2 (Experimental)
  Interventions: Other: Education Program Type 2

INTERVENTIONS:
Other: Education Program Type 1 — The first part of the education program involves four weeks of in-person classes (2 hours per class) given once per week with homework assignments of approximately 30 minutes per day for at least 5 days per week. The second part of the education program involves home-based activities only, performed approximately 30 minutes per day for at least 5 days per week.
  Arms: Education Program Type 1
Other: Education Program Type 2 — The first part of the education program involves four weeks of in-person classes (2 hours per class) given once per week with homework assignments of approximately 30 minutes per day for at least 5 days per week. The second part of the education program involves home-based activities only, performed approximately 30 minutes per day for at least 5 days per week.
  Arms: Education Program Type 2

SUMMARY:
Chronic pain (pain that is that is present for a long period of time) is very common among people with spinal cord injury (SCI). Unfortunately, chronic pain is very difficult to treat. Many treatments reduce chronic pain only partially. As a result, many people with SCI must find ways of accomplishing daily activities even though they have pain.

The purpose of this research study is to determine how well two different kinds of education programs reduce the extent to which chronic pain interferes with daily life and well-being.

DETAILED DESCRIPTION:
Pain is a highly prevalent and disabling condition among persons with spinal cord injury (SCI). Unfortunately, current pain treatments offer incomplete relief, produce side effects, and/or involve significant cost. Low-risk, low-cost treatments capable of addressing residual pain and pain-related disability are greatly needed. A number of research studies have associated educational interventions with improvements in pain-related outcomes.

The overall goal of the proposed pilot study is to evaluate the feasibility, acceptability, and potential benefits of two types of educational programs for people with chronic pain and spinal cord injury. This study aims to identify a low-cost, low-risk treatment option that empowers people with pain and SCI to improve their functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury for at least one year
* Chronic pain for at least three months that is moderate to severe (rated at or above 4/10 on a scale of 0 to 10 where 0 = "no pain" and 10 = "pain as bad as you can imagine")
* Fluent in English
* Not currently starting a new pain treatment or changing a previous pain treatment

Exclusion Criteria:

* Cancer or conditions that may worsen over time (such as multiple sclerosis, Parkinson Disease, Alzheimer's disease) and may affect my physical or mental functioning
* Significant difficulties with learning or memory
* Previous participation in a health and function education program specifically designed for people with chronic pain and SCI
* Inability to understand English
* Presence of other conditions not related to SCI that cause pain (such as fibromyalgia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain interference with activities | Week 10 versus baseline
  The extent to which pain interferes with daily activities will be measured with the Life Interference Subscale of the Multidimensional Pain Inventory (MPI-LIS). The MPI-LIS is a 10-item self-report of extent of interference of pain with life activities and the enjoyment of life. The subscale will be modified to remove two items related to work, as recommended based on a factor analysis of the subscale in persons with SCI.

SECONDARY OUTCOMES:
Pain intensity | Week 10 versus baseline
  Pain intensity will be rated on a 0-10 numerical rating scale (0="no pain" and 10="pain as bad as you can imagine").
Mental health and well-being | Week 10 versus baseline
  The Brief Patient Health Questionnaire and Perceived Stress Scale will be used to assess changes in mental health that occur between baseline and the end of the education program.
Pain attitudes | Week 10 versus baseline
  The Survey of Pain Attitudes will be used to assess changes in thoughts and beliefs about pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Zanca, PhD, MPT, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

REFERENCES:
- See also: Kessler Foundation Home Page — http://KesslerFoundation.org